CLINICAL TRIAL: NCT06387277
Title: Assessment of the Impact of Skin Microbiota on Wound Healing Process Using an Epidermally Ablated Skin Model of Erbium YAG Laser by Comparing Areas Treated With RV1551P GB3224 With Untreated: Exploratory Study
Brief Title: Re-epithelialization Efficacy Evaluation of Cosmetic Product RV1551P vs Non-treated Forearm of Healthy Adult Women
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV1551P20220376
Record Dates: First submitted 2024-04-09; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Female; 20 to 45 years old; re-epithelialization; microbiota; metabolomic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Swab samples on the skin surface to access skin microbiota and metabolites produced by the skin and microbiota.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Arms of healthy female from 20 to 45 years old: It is a randomized intra-individual comparative study where two areas of the skin are ablated using an erbium YAG laser at Visit 1, with a surface area of approximately 6cm² (Z1 and Z3). Additionally, two healthy areas (Z2 and Z4), with a similar surface area, are identified on each forearm. The study involves comparing the areas treated with the product RV1551P GB3224 to the untreated areas (randomized arms).
  Interventions: Other: RV1551P GB3224

INTERVENTIONS:
Other: RV1551P GB3224 — RV1551P GB3224 Approximately 2 mg/cm² of product is applied to the Z1 or Z3 study areas (randomization).
  From D1 to D2, a single product application is done at the study center by the subject in the presence of the clinical research technician (CRT) after epidermal ablation with an erbium YAG laser. After application, a dressing is placed on the measurement area and removed the following day at the center on D2 and D3 by the CRT before measurements.
  From D3 to D18, two product applications are done with a minimum 4-hour interval:
  * On visit days (D3, D5, D8, D10, D12, D15): an application is done at the study center by the subject in the presence of the CRT after measurements. A second application is done at home in the evening.
  * On non-visit days (D4, D6, D7, D9, D11, D13, D14, D16, D17, D18): the subject applies 2 product applications at home (morning and evening).
  Subjects receive the product at the end of visit 3 and return it at the last visit (visit 9).

SUMMARY:
The aim of this study was to evaluate the impact of the product RV1551P GB3224 on skin microbiota during wound healing process, based on swab samples collected from lesion areas using an epidermally ablated skin model of erbium YAG laser.

DETAILED DESCRIPTION:
This study is a monocentric, open-label, intra-individual, controlled and randomized study conducted in 21 healthy adults.

A comparison is done between areas treated with the product RV1551P GB3224 and untreated areas (randomized arms).

The swab samples are performed on 4 study areas: 2 areas on the volar aspect of each forearm identified Z1, Z2, Z3 and Z4. Two areas are epidermally ablated with an erbium YAG laser at Visit 1 (D1) with a surface around 6cm² (Z1 and Z3): one area is treated with the product RV1551P GB3224 and the other one is untreated. On these areas, four swab samples are performed: at Day 1 before and after the laser act at the inclusion visit (V1-D1), at Day 5 (V4-D5), at visit corresponding to complete wound healing (re-epithelialization time) and at the end of study (V9-D19).

Two healthy areas (Z2 and Z4), with a surface around 6cm², are identified on each forearm. One of these areas is treated with the product RV1551P GB3224. On these areas, two swab samples are performed: at the inclusion visit (V1-D1), and at the end of study (V9-D19).

ELIGIBILITY:
Inclusion Criteria:

1. Criteria related to the population:

   * Male or female, from 20 to 45 years old included.
   * Phototype I, II or III according to the Fitzpatrick classification.
   * Subject smoking ≤ 10 cigarettes / day containing nicotine, paper and/or electronic cigarette equivalent.
   * Subject agreeing not to expose his forearms to UV (natural or artificial) throughout the duration of the study and up to 3 months after the end of participation in the study.
   * If the subject is a woman of childbearing age:

     i. Subject who used an effective method of contraception, evaluated by the investigator for at least 8 weeks before inclusion in the study.

   ii. Subject agreeing to continue using it during all the study and up to 5 days after the last products application, in order to avoid pregnancy during exposure to the study products.
   * Absence from participation in a clinical research protocol.
   * Signature of the informed consent form.
   * Affiliation to social security scheme or beneficiary of such a scheme.
2. Criteria related to treatment:

   * Subject protected by a tetanus vaccination according to the vaccination schedule established by the Public Health Agency.

Exclusion Criteria:

1. Criteria related to the population:

   * Pregnancy or breastfeeding ongoing or planned during the study.
   * Subject deprived of freedom through a legal or administrative decision, or in care or under legal guardianship.
   * Subject unable to comply with the requirements of the protocol according to the opinion of the investigator.
   * Physical or linguistic impairment for signing the informed consent form.
   * Current participation planned participation or participation in previous weeks or months in another clinical study that may interfere with the study according to the opinion of the investigator.
   * Subject who has participated twice in a clinical study using the Er YAG laser on the forearms.
2. Criteria related to diseases and general health:

   * Subject with known immunodeficiency.
   * Subject with known acquired immunodeficiency syndrome.
   * Subject with known infectious hepatitis or a known history of hepatitis B or C.
   * Subject with a known history of allergy or contact dermatitis induced in particular by the latex, the plaster, the local anesthetic, the local antiseptic or one of the components of the study products.
   * Subject with a recognized addiction to alcoholism or drug.
   * Subject having already presented cicatrization disorders.
   * Subject presenting pathology of cicatrization or pathology with consequences on cicatrization such as diabetes.
   * Subject with a disease including skin disease in progress on the upper limbs that may interfere with the interpretation of the evaluation criteria according to the opinion of the investigator.
   * Subject with a history of atopic eczema on the upper limbs (arms, forearms, hands).
   * Subject with skin lesion, solar erythema, tanning marks, scar(s), tattoo(s), significant hair growth, nevus, visible or prominent veins on study areas that may interfere with the interpretation of the evaluation criteria according to the opinion of the investigator.
   * Subject presenting hereditary disorders or acquired haemostasis.
   * Subject with congenital methemoglobinemia or porphyria.
   * Subject with chronic or acute pathology able to interfere with the results of the study according to the opinion of the investigator.
3. Criteria related to treatments

   * Diuretic or diuretic systemic treatment initiated or modified in the 2 months prior to the inclusion visit or started at the inclusion visit or whose start is scheduled during the study.
   * Treatment liable to induce methemoglobinemia (sulfonamides, dapsone, metoclopramide, flutamide, sodium nitroprusside) in the 14 days prior to the inclusion visit or during the inclusion visit.
   * Systemic corticosteroid treatment in the 14 days prior to the inclusion visit or ongoing during the inclusion visit or planned during the study.
   * Systemic treatment that may affect haemostasis, including anti-coagulant, antiplatelet therapy, within 7 days prior to the inclusion visit or ongoing at the inclusion visit or planned during the study.
   * Systemic treatment with non-steroidal anti-inflammatory drug in the 7 days prior to the inclusion visit or ongoing at the inclusion visit (from 3 days of intake).
   * Systemic treatment liable to affect the healing process according to the opinion of the investigator in the weeks prior to the inclusion visit, ongoing at the inclusion visit or planned during the study.
   * Systemic or topical antibiotic and/or antifungal treatment within 4 weeks prior to the inclusion visit or ongoing at the inclusion visit.
   * Topical antiseptic treatment applied to the upper limbs (including the hands) within 2 weeks prior to the inclusion visit or ongoing at the inclusion visit.
   * Topical non-steroidal anti-inflammatory treatment, topical corticosteroids, immunomodulators applied to the upper limbs (including the hands) in the 15 days prior to the inclusion visit or ongoing at the inclusion visit or planned during the study.
   * Physical treatment including forearm radiotherapy on the forearm in the 6 months prior to the inclusion visit or ongoing at the inclusion visit or planned during the study.
   * Phototherapy treatment on the forearm in the 8 weeks prior to the inclusion visit, ongoing at the inclusion visit or planned during the study.
   * Subject with intense and prolonged exposure to UV (natural or artificial) in the forearms in the 2 weeks prior to the inclusion visit or planned during the study.
   * Any other treatments taken, applied or modified in the weeks prior to the inclusion visit, ongoing at the inclusion visit or planned during the study that may interfere with the study according to the opinion of the investigator.
   * Use of keratolytic, exfoliating or self-tanning products on the upper limbs (including hands) in the 14 days prior to the inclusion visit or on the day of the inclusion visit.
   * Use of a skin care product on the upper limbs (including the hands) in the 7 days prior to the inclusion visit or the day of the inclusion visit.
   * Application of water, hygiene products on the upper limbs in the 8 hours prior to the inclusion visit, without hygiene usual routine modification during the study.
   * Subject having modified his usual body hygiene routine the day before the inclusion visit or planned to modify during the study.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Subjects have been recruited from the panel of the centre. An investigator made a dermatological examination of the subjects before inscription in the panel.
  Data from this clinical examination, stored in the computer database with the consent of the subjects, can ensure the recruitment; computer software being questioned based on the eligibility criteria of the study.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Time to re-epithelialization as assessed by in vivo examination by the investigator and standardized photographs taken with a C Cube Camera® | Change from baseline to 10 minutes after the YAG laser act, before the application of the product. During the following visits (Day 3, Day 5, Day 8, Day 10, Day 12, Day 15, Day 19), the photographs will be taken before the product is applied.
  The wound disappearance is assessed by the investigator from in vivo examination and from standardized photographs of the study areas taken at each visit with a C Cube Camera®. Illustrative photographs will be collected by NomadCam©

SECONDARY OUTCOMES:
Skin microbiota diversity from swab samples. | Change from baseline to 10 minutes after the YAG laser act, Day 5, re-epithelialization time and Day 19, before the application of the product.
  Microbiota composition is analyzed by 16S and ITS1sequencing.
Skin microbiota composition from swab samples. | Change from baseline to 10 minutes after the YAG laser act, Day 5, re-epithelialization time and Day 19, before the application of the product.
  Shannon, Chao1 and Observed diversity indexes for bacteria and fungi are calculated with the number of identified sequences obtained with 16S and ITS1sequencing.
Metabolomic analysis from swab samples | Change from baseline to 10 minutes after the YAG laser act, Day 5, re-epithelialization time and Day 19, before the application of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer THEUNIS, MD, Principal Investigator — SKIN RESEARCH CENTRE - Toulouse
Locations (1):
- Skin Research Centre, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No